CLINICAL TRIAL: NCT06111664
Title: Anergia-anhedonia by Lithium-induced Phosphorus Diabetes
Acronym: ALIPo-D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8953
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Mood Disorders
Keywords: Diabetes, Phosphate; Anergia-anhedonia; Lithium (Li+); Mood Disorders
MeSH Terms: conditions — Mood Disorders; Hypophosphatemia, Familial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lithium (Li+) is prescribed to 1‰ of the French population (~ 60,000 patients). More than half of patients describe subjective symptoms linked to Li+ (SSL) similar to those of chronic fatigue syndrome: muscle weakness, fatigability, cognitive disorders, emotional blunting. SSL are the 2nd cause of stopping Li+ (28%), just behind kidney problems (30%).

In animals, the administration of lithium (Li+) increases the urinary excretion of phosphate (Pi) by 6, inducing phosphate diabetes (DPi). However, idiopathic forms of DPi explain up to 10-15% of chronic fatigue syndromes and these disappear when supplementing with Pi (± vitamin D).

In humans, the introduction of Li+ leads to a reduction in serum phosphate but we have not found any publication on the possible induction of DPi or on a possible link between DPi and SSL.

However, the dosages necessary to detect a DPi are carried out during the annual follow-up assessment of patients on Li+. All you have to do is calculate the standardized maximum reabsorption rate of Pi (TmPi) to make the diagnosis! Finally, if the patients presenting with DPi turn out to be the same as those who complain of SSL, we can imagine that correcting the first by simple supplementation with Pi (± vitamin D) could provide relief.

DETAILED DESCRIPTION:
The aim of the study is to determine the prevalence of hypophosphatemia, DPi and SSL in a population of ambulatory patients controlled on Li+ (> 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥ 18 years old)
* Man or woman
* Subject balanced on Li+ (> 6 months, regardless of the underlying pathology).
* Outpatient monitoring by one of the members of CEDRA (Alsace expert center for resistant depression).
* Subject not opposing, after information, the reuse of their data for the purposes of this research

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Subject under judicial protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) balanced on Li+ (> 6 months, regardless of the underlying pathology).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04-24 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypophosphatemia, DPi and SSL at the population level. | from 6 months after lithium treatment (Li+)
  The prevalence is determined retrospectively on a population balanced on lithium (Li+) for more than 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- CENTRE DE NEUROMODULATION NON INVASIVE DE STRASBOURG (CEMNIS) - CHU de Strasbourg - France, Strasbourg, France